CLINICAL TRIAL: NCT06769490
Title: Phase 1 Dose Escalation and Expansion of Ziftomenib in Combination With Quizartinib in Acute Myeloid Leukemia
Brief Title: Dose Escalation and Expansion of Ziftomenib in Combination With Quizartinib in Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1193; NCI-2024-10248 (Other: NCI-CTRP Clinical Trials Registry); NCI-2025-00080 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ziftoenib + Quizartinib Q4W (Experimental): Participants will be randomized to study
  Interventions: Drug: Ziftomenib; Drug: Quizartinib

INTERVENTIONS:
Drug: Ziftomenib — Participants will receive treatment in tablet form
Drug: Quizartinib — Participants will receive treatment in tablet form

SUMMARY:
The goal of this all-oral combination is to deliver safe and effective therapy for the largest portion of AML subtypes (NPM1mt, KMT2Ar, NUP98r ~ 40-45%).

DETAILED DESCRIPTION:
Primary Objective:

Cohort 1A: To determine the recommended phase 2 dose (RP2D) of ziftomenib in combination with quizartinib and assess the safety and the maximum tolerated dose (MTD).

Secondary Objectives:

To assess the preliminary efficacy of the combination of quizartinib and ziftomenib by FLT3 mutational status.

To assess overall survival (OS), relapse-free survival (RFS), event-free survival (EFS) and duration of response (DOR).

To characterize the pharmacokinetic profile of ziftomenib and quizartinib when used in combination.

To assess minimal residual disease negativity by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. Age . 18 years.
2. ECOG performance status of < 2.
3. Relapsed or refractory AML or myeloid mixed-phenotype acute leukemia (MPAL) with NPM1mt, or KMT2Ar, or NUP98r.
4. WBC must be below 25,000/ ƒÊL at time of enrollment. Patients may receive cytoreduction prior to enrollment.
5. Baseline ejection fraction must be > 40%.
6. Adequate hepatic function (total bilirubin < 2x upper limit of normal (ULN) unless increase is due leukemic involvement (<2.5 ULN), unless due to ongoing hemolysis or Gilbert's syndrome and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
7. Adequate renal function with an estimated glomerular filtration rate . 50 mL/min (using Cockcroft-Gault) unless related to disease.
8. Able to swallow pills.
9. Patient or parent/guardian is willing and able to provide informed consent.
10. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy, whichever is longer. Oral hydroxyurea and/or cytarabine (up to 1 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI.

    Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
11. Women of childbearing potential must agree to adequate methods of contraception during the study and at least 7 months for females and 4 months for males after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and at least 4 months after the last treatment.

Exclusion Criteria:

1. Prior treatment with a menin inhibitor.
2. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
3. Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
4. Patients with a concurrent active malignancy under treatment.
5. Known active hepatitis B (HBV) or Hepatitis C (HCV) or HIV infection.
6. Female subjects who are pregnant or breast-feeding.
7. Patient has an active uncontrolled infection.
8. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class .II), life-threatening, uncontrolled arrhythmia including ventricular arrythmias or torsades de pointes, cerebrovascular accident, or transient ischemic attack.
9. History of sustained bradycardia of less than 50 beats per minute unless the subject has a pacemaker.
10. Diagnosis of or suspicion of congenital long QT syndrome (including family history of congenital long QT syndrome).
11. Uncontrolled hypertension with a systolic blood pressure .180 mmHg or diastolic blood pressure .110 mmHg, sustained despite optimal medical management.
12. QTc >450 msec using the Fridericia Formula.
13. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate. Patients under legal protection measure (guardianship, trusteeship or safeguard of justice) and/or uncontrolled psychiatric comorbidities, ongoing illicit substance abuse, inability, any impairment or unwillingness to comply with the treatments, follow-up, requirements and procedures of this clinical trial.
14. Clinically active central nervous system (CNS) leukemia.
15. Patients with Grade > 2 active acute GVHD, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2030-09-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org